CLINICAL TRIAL: NCT04249700
Title: Investigating the Effect of Single-session Sauna Use on Body Temperature
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Mount Zion Health Fund (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: HEATBED1
Record Dates: First submitted 2020-01-23; First posted 2020-01-31 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Core Body Temperature 101.3 F

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Whole-body Hyperthermia (WBH) (Experimental): All participants receive WBH for 80-110 minutes in the Curve Sauna Dome infrared sauna. Participants lay supine in the sauna during this time, and their head is external to the sauna.
  Interventions: Device: Curve Sauna Dome

INTERVENTIONS:
Device: Curve Sauna Dome — All participants receive WBH for 80-110 minutes in an infrared sauna. Participants lay supine in the sauna during this time, and their head is external to the sauna.

SUMMARY:
Whole-body hyperthermia (WBH) to an internal temperature of 38.5 C (101.3 F) using an infrared heating device has been associated with significant reductions in clinical depression. This prior work utilized a WBH medical device that is manufactured in Germany, is not FDA approved, and is not widely available. The goal of this initial pilot project is to ascertain whether an infrared sauna, the Curve Sauna Dome, which is readily accessible (i.e., can be purchased by consumers in the US) can be used to conduct WBH that achieves an internal body temperature of of 101.3 F in healthy volunteers.

DETAILED DESCRIPTION:
Prior work has demonstrated that whole body hyperthermia (WBH) to an internal temperature of 38.5 C (101.3 F) using an infrared heating device is associated with significant reductions in clinical depression. This prior work utilized a Heckel WBH device, a medical device manufactured in Germany that is not FDA-approved and that is not widely available. The goal of this pilot project is to ascertain whether the Curve Sauna Dome, an infrared sauna that is readily accessible (i.e., can be purchased by consumers in the US) can be used to conduct WBH that achieves an internal body temperature of of 38.5 C (101.3 F) in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Male or pre-menopausal female volunteers aged 18-45.
* Able to understand the nature of the study and able to provide written informed consent prior to conduct of any study procedures.
* Able to communicate in English with study personnel.
* Able to lay supine for 2 hours in a sauna.
* BMI <=30
* Waist size of <=40 inches for men or <=35 inches for women
* Have a smartphone
* If female, and sexually active with men, must agree to use non-hormonal birth control (e.g., barrier methods, partner with vasectomy, tubes tied, copper IUD)
* Must have negative pregnancy test day of sauna session

Exclusion Criteria:

* Any history of or current mental health condition
* Any current medical condition requiring medical treatment
* Any history or current substance misuse/abuse
* Regular use of any nicotine products, including cigarettes, e-cigarettes, chewing tobacco, or other forms of nicotine
* Unable to refrain from psychoactive dietary or herbal products, including marijuana, in the 2 weeks prior to study participation
* Breastfeeding or pregnant women, women intending to become pregnant within 6 months of the screening visit
* Sexually active women of child bearing potential who are not using a medically accepted physical means of contraception (defined as non-hormone-based implant, condom, diaphragm, status-post tubal ligation, or partner with vasectomy)
* Current use of hormone-based birth control, such as IUD or oral contraceptive
* Needing to use of any medication that might impact thermoregulatory capacity within 5 days of the sauna session, including: stimulants, diuretics, barbiturates, beta-blockers, antipsychotic agents, anti-cholinergic agents or chronic use of antihistamines, aspirin (other than low-dose aspirin for prophylactic purposes), non-steroidal anti-inflammatory drugs (NSAIDs), systemic corticosteroids, cytokine antagonists
* Current antidepressant medications (all classes) or use within the past 30 days

The following medications in these timeframes:

* Antibiotics (past 60 days)
* Pain medication (opioids) due to procedure, e.g., dental procedure (past 30 days)
* Emergency contraception pill (past 60 days)
* Benzodiazepines, e.g., procedure (past 30 days)
* Use of any other medication that in the judgment of the PI would increase risk of study participation or introduce excessive variance into physiological or behavioral responses to WBH
* Known hypersensitivity to infrared heat exposure
* Unwilling to refrain from sauna use outside of study procedures for one week before and one week after sauna session

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2019-09-13 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Sauna Curve Dome successfully induces a core body temperature of 101.3 | Duration of time in Curve Sauna Dome, up to ~110 minutes
  Achieving core body temperature of 101.3 F using a rectal temperature assessment method
Adverse Events Causing Cessation of Curve Sauna Dome Session | Duration of time in Curve Sauna Dome, up to ~110 minutes
  Any adverse event causing stopping of sauna session prior to achieving 101.3 F

SECONDARY OUTCOMES:
Time to Achieve Core Body Temperature of 101.3 F in Curve Sauna Dome | Duration of time in Curve Sauna Dome, up to ~110 minutes
  Amount of time before participant achieves core body temperature of 101.3 F using a rectal temperature assessment method

CONTACTS AND LOCATIONS:
Overall Officials: Ashley E Mason, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
This is currently a feasibility test to ascertain if the procedure can attain the desired outcome. Results will be published.

REFERENCES:
- [Result] Mason AE, Fisher SM, Chowdhary A, Guvva E, Veasna D, Floyd E, Fender SB, Raison C. Feasibility and acceptability of a Whole-Body hyperthermia (WBH) protocol. Int J Hyperthermia. 2021;38(1):1529-1535. doi: 10.1080/02656736.2021.1991010. PMID 34674592